CLINICAL TRIAL: NCT02814487
Title: A Pilot Validation Study Comparing "DAM" a Smartphone Application With the Composite MSFC Score Intra-individually Among Multiple Sclerosis Patients
Brief Title: MSFC Versus DAM. A Smartphone Application for Multiple Sclerosis Self-assessment.
Acronym: DAM
Status: Completed | Type: Observational
Sponsor: Ad scientiam (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Other Study IDs: P003
Record Dates: First submitted 2016-06-22; First posted 2016-06-27 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-06

CONDITIONS: Multiple Sclerosis
Keywords: DAM; multiple sclerosis; MSFC; application; smartphone
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Multiple Sclerosis Functional Composite score (MSFC) is one of the gold standard for multiple sclerosis (MS) patient clinical evaluation. However, its practical implementation is not always optimal as it can prove to be very time consuming. Moreover, it often constrains the range of tests used and is not a particularly good marker for patient real life disability status.

A mobile application called Digital Self-Assessment for Multiple Sclerosis (DAM) was developed in order to replicate each of MSFC tests available in order to assess MS progression in the patient environment.

DETAILED DESCRIPTION:
Patients are selected during a consultation at the Neurology department of the Pitié-Salpêtrière Hospital (France). Each patient is given access to DAM on their own or a provided iPhone. During the enrolment visit, patients have to complete a MSFC and DAM evaluation (V0). Through a push-notification on their phone, patients are reminded to perform two DAM evaluations at home at days 30 (V1) and 60 (V2). At day 90 (V3), they have to come back to hospital for a second MSFC and DAM evaluation

ELIGIBILITY:
Inclusion Criteria:

* Patients with an established diagnosis of Multiple sclerosis according to the MacDonald criterias whatever the progression stage, that are monitored by Dr. Maillart as part of her consultation at the Neurology department of the Pitié-Salpêtrière Hospital.
* Patients with an iPhone (at iOS 8 or higher).
* Patients age ≥18 years.
* Patients with an initial score of EDSS between 0 to 6.5
* No attack since at least 1 month
* Last Solumedrol injection at least 1 month ago

Exclusion Criteria:

* Patients who are not capable of using a smartphone application.
* Patients who do not have the capacity to give their consent.
* Patients who do not speak French
* Patients who are bedridden or with a daily activity of less than 2 hours per day
* Patients with acute asthenia
* Patients experiencing an attack once enrolled in the study (will be considered as dropouts)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with multiple sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-12; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
correlation between the MSFC score and the DAM score | At Day 0

SECONDARY OUTCOMES:
correlation between the DAM score | At Day 0 and Day 30
correlation between the DAM score | At Day 60 and Day 90
correlation between the the MSFC and the DAM score | At Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth MAILLARD, MD, Principal Investigator — Pitié Salpêtrière Hospital, Paris

IPD SHARING:
Plan to Share IPD: No